CLINICAL TRIAL: NCT04687410
Title: Randomized Comparison of Tissue Quality and Molecular Yield Between a Novel Crown-cut Biopsy Needle (FNB) and a Standard Aspiration Needle (FNA) for EUS Guided Diagnosis of Solid Pancreatic Lesions
Brief Title: Novel Crown-cut Biopsy Needle (FNB) vs Standard Aspiration Needle (FNA) for EUS-guided Diagnosis of SPLs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter Vilmann MD, DSc, HC, FASGE (Other)
Collaborators: Hvidovre University Hospital (Other); Department of Gastroenterology, Ponderas Academic Hospital Bucharest, Romania (Unknown); Endoscopy Unit, Odense Hospital, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Peter Vilmann MD, DSc, HC, FASGE, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: H-20006798
Record Dates: First submitted 2020-06-22; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Pancreas Neoplasm; Pancreas Cancer
Keywords: fine needle aspiration; fine needle biopsy; solid pancreatic lesion; pancreatic neoplasm; pancreatic cancer; endoscopic ultrasound; EUS-FNA; EUS-FNB
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FNA (Active Comparator)
  Interventions: Device: ProControl, MediGlobe
- FNB (Experimental)
  Interventions: Device: TopGain, Medi-Globe

INTERVENTIONS:
Device: ProControl, MediGlobe — standard 22G FNA needle
  Arms: FNA
Device: TopGain, Medi-Globe — novel 22G crown-cut FNB needle
  Arms: FNB

SUMMARY:
The aim of this study is to compare tissue quality and molecular yield between a novel crown-cut biopsy needle (FNB) and a standard aspiration needle (FNA) for EUS-guided diagnosis of solid pancreatic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a newly discovered SPL scheduled for EUS-guided tissue acquisition who can understand and provide a written consent.

Exclusion Criteria:

* Patients with uncorrected coagulopathies (INR >1.5 or platelet count <50,000) or patients treated with anticoagulants that cannot be discontinued.
* Pregnant or lactating females.
* Interposed, large vessels between the transducer and the target lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Amount of tissue micro-fragments | 1 month
  Comparison of median number of tissue micro-fragments
Diagnostic tissue area | 1 month
  Comparison of total diagnostic tissue area in um2
Total tissue area | 1 month
  Comparison of total total tissue area in um2

SECONDARY OUTCOMES:
Diagnostic yield | 1 month
  diagnostic yield - defined by percentage of diagnostic samples in each group
Diagnostic performance | 12 month
  Sensitivity and specificity, where final diagnosis is either established by subsequent histopathological confirmation or other evidence (clinical, radiological) of malignant disease at a minimum of 12 months of follow-up
Adverse event rate | 1 month
  Comparison of proportions of patients experiencing AE in each group as defined by ASGE's lexicon on adverse events in endoscopy
Mean DNA concentration | 6 months
Suitability for molecular analyses | 6 months
  Percentage of samples where NGS analysis was successful

CONTACTS AND LOCATIONS:
Locations (1):
- Gastro Unit, Division of Endoscopy, Herlev, Danmark, Denmark